CLINICAL TRIAL: NCT00263185
Title: A Double-Blind, Randomized, Placebo Controlled Trial of High Dose Vitamin D Therapy On Musculoskeletal Symptoms and Bone Mineral Density in Anastrozole-Treated Early Stage Breast Cancer Patients With Marginal Vitamin D Status
Brief Title: High Dose Vit D Musculoskeletal Symptoms & Bone Density in Anastrozole-Treated Breast Cancer With Marginal Vit D Status
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 05-0498 / 201012921
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Vitamin D; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Treatment Group (Experimental): Patients with baseline 25OH vitamin D level of 10-19 ng/ml.
  * Calcium carbonate 1000 mg/day
  * Vitamin D 400 units daily.
  * Vitamin 50,000 IU/wk x 16 weeks and then once a month for a total of 6 months.
  Patients with baseline 25OH vitamin D level of 20-29 ng/ml.
  * Calcium carbonate 1000 mg/day
  * Vitamin D 400 units daily.
  * Vitamin 50,000 IU/wk x 8 weeks and then once a month for a total of 6 months.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Calcium carbonate; Drug: Vitamin D
- Control Group (Placebo Comparator): Patients with baseline 25OH vitamin D level of 10-19 ng/ml.
  * Calcium carbonate 1000 mg/day
  * Vitamin D 400 units daily.
  * Placebo once per week x 16 weeks and then once a month for a total of 6 months.
  Patients with baseline 25OH vitamin D level of 20-29 ng/ml.
  * Calcium carbonate 1000 mg/day
  * Vitamin D 400 units daily.
  * Placebo once per week x 8 weeks and then once a month for a total of 6 months.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Calcium carbonate; Other: Placebo
- Observational Group (Other): Patients with a baseline Vitamin D level below 10 ng/ml.
  * Calcium carbonate 1000 mg/day
  * Vitamin D 400 units daily.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Dietary Supplement: Vitamin D
Dietary Supplement: Calcium carbonate
Drug: Vitamin D
  Arms: Active Treatment Group
Other: Placebo
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether Vitamin D supplementation reduces the symptoms of muscle stiffness and joint tenderness that some patients may develop after starting therapy with Anastrozole for breast cancer.

DETAILED DESCRIPTION:
This is a pilot, double-blind, randomized, placebo-controlled study with the following aims:

* To compare the effects of high dose vitamin D versus standard dose vitamin D on musculoskeletal pain in breast cancer patients receiving anastrozole when vitamin D levels are in the insufficient but not deficient range (10 to 29 ng/ml).
* To evaluate the prevalence of vitamin D insufficiency/deficiency in post-menopausal women with a history of breast cancer who are treated with anastrozole and have musculoskeletal symptoms versus those who are asymptomatic.
* To establish correlations between levels of vitamin D, the levels of PTH, the degree of bone loss and the severity of musculoskeletal symptoms.
* To evaluate the effect of standard dose versus high dose Vitamin D replacement on bone density in post-menopausal women with a history of breast cancer who are treated with anastrozole and have musculoskeletal symptoms.

ELIGIBILITY:
Inclusion Criteria

* Women with a diagnosis of hormone receptor positive invasive breast cancer (Stage I-IIIB) or ductal carcinoma in situ (DCIS)
* Postmenopausal status
* Completed at least 8 weeks of anastrozole as adjuvant therapy prior to study entry
* Completed systemic chemotherapy and radiation treatments when indicated
* Serum Calcium ≤ 10.3 mg/dL
* Patients with marginal 25 OH Vitamin D level (between 10 and 29 ng/ml) will be in the Randomized Group or Low 25 OH Vitamin D level (less than 10 ng/ml) will be in Observational Group
* 24-hour urine Calcium excretion ≤ 250 mg/g (calculated by dividing 24 hour calcium by 24 hour creatinine)
* A history of generalized musculoskeletal pain with or without localized regions or discomfort that has developed or worsened since starting adjuvant aromatase inhibitor therapy

Exclusion Criteria

* Known metastatic disease
* History of kidney stones
* History of active primary hyperparathyroidism
* History of Paget's disease of the bone
* History of severe arthritis, rheumatoid arthritis, or severe neuropathy
* Normal 25 OH Vitamin D level (≥ 30 ng/ml)
* Medical or psychiatric condition which may preclude protocol compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To compare the effects of high dose vitamin D versus standard dose vitamin D on musculoskeletal pain in breast cancer patients receiving anastrozole when vitamin D levels are in the insufficient but not deficient range (10 to 29 ng/ml). | 6 months for randomized phase, 12 months for open-label phase

SECONDARY OUTCOMES:
To evaluate the prevalence of vitamin D insufficiency/deficiency in post-menopausal women with a history of breast cancer who are treated with anastrozole and have musculoskeletal symptoms versus those who are asymptomatic. | 6 months for randomized phase, 12 months for open-label phase
To establish correlations between levels of vitamin D, the levels of PTH, the degree of bone loss and the severity of musculoskeletal symptoms. | 6 months
To evaluate the effect of standard dose versus high dose Vitamin D replacement on bone density in post-menopausal women with a history of breast cancer who are treated with anastrozole and have musculoskeletal symptoms. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Rastelli, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu